CLINICAL TRIAL: NCT00483860
Title: A Phase I Study of Oral Topotecan in Subjects With Cancer and Impaired Renal Function
Brief Title: A Phase I Topotecan Study in Subjects With Cancer and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKF104864/722
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Solid Tumours
Keywords: Cancer; Solid tumor,; normal renal function; renal impairment,; prior platinum-based chemotherapy,
MeSH Terms: conditions — Neoplasms; Renal Insufficiency | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topotecan (Experimental): once a day
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Topotecan — once a day

SUMMARY:
To determine the effect of renal impairment and prior platinum-based chemotherapy on the safety and blood levels of topotecan administered orally

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
2. Age 18 years or older.
3. A performance status score of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) Scale.
4. Histologically- or cytologically-confirmed advanced solid tumors.
5. Failed conventional therapy for their tumor type; or subjects who have a tumor type for which no standard effective therapy exists; or subjects for whom single-agent topotecan therapy is suitable.
6. Completion of a 24-hour urine collection within 14 days prior to the first dose to calculate the creatinine clearance value and determine the renal impairment category (refer to Appendix 8).
7. Using Cockcroft-Gault formula (refer to Appendix 6), documentation of stable renal function should be performed within 14 days of the first scheduled dose of study medication using at least 2 serum creatinine values separated by a minimum of 7 days. Stable renal function is defined as:

   1. ≤25% change for CrCl <40 mL/min or
   2. ≤10 mL/min change for CrCl ≥40 mL/min NOTE: Documentation of stable renal function will NOT be required if the 24-hour urine collection to determine the renal impairment category is completed within 7 days prior to the first dose.

Exclusion Criteria:

* Currently undergoing dialysis.
* Pregnant or lactating.
* Women of childbearing potential who refuse to either abstain from sexual intercourse or practice adequate contraception
* Male subjects with female partners of childbearing potential who have not had a prior vasectomy or if both the male subject and the female partner refuse to use adequate contraception beginning 14 days before exposure to study drug, continuing throughout the clinical trial, and for a period of 3 months after the last dose of study drug.
* Uncontrolled emesis, regardless of etiology.
* Bilirubin > 1.5 X ULN.
* SGOT/AST, SGPT/ALT and alkaline phosphatase >2 times the upper limit of normal (ULN) if no evidence of potentially associated metastases (e.g., liver or bone) by computed tomography (CT) or magnetic resonance imaging (MRI). If potentially associated metastases (e.g., liver or bone) are present, subjects with <5 times ULN are eligible to participate, following discussion with and approval from a GSK Medical Monitor.

Hematological values outside of acceptable ranges. Active infection. Prior anti-cancer therapy, including, but not limited to, chemotherapy (except nitrosurea or mitomycin C), radiotherapy, biologic therapy, investigational therapy or major surgery within 21 days of the first scheduled dose of study drug. Prior nitrosurea of mitomycin C chemotherapy within 6 weeks of first scheduled dose of study drug. Failure to recover to Grade 1 or better from any toxicity (except alopecia) related to prior anti-cancer therapy by Day 1, Course 1 unless agreed to by a GSK Medical Monitor and the Investigator. Clinical evidence of a gastrointestinal (GI) condition (i.e., removal of a portion of the stomach, recent GI obstruction or GI neuropathy) or taking drugs that would alter GI absorption or motility. Currently taking or will require treatment with cyclosporin A. Concurrent severe medical problems unrelated to the malignancy, which would significantly limit full compliance with the study or expose the subject to extreme risk (including major surgery within 21 days or placement of biliary stents or nephrostomy tubes within 7 days). History of allergic reactions to topotecan or compounds chemically related to topotecan (e.g., irinotecan).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-06-20 (Actual); Primary Completion 2012-02-06 (Actual); Study Completion 2012-02-06 (Actual)

PRIMARY OUTCOMES:
Comparison of blood levels of topotecan following oral and IV dosing; | blood samples will be drawn on Day 1 and Day 8 of Courses 1 and 2.

SECONDARY OUTCOMES:
Assessment of clinical laboratory tests, cardiac monitoring and disease progression. Comparison of blood levels of topotecan when taken orally with and without food; | blood samples will be drawn on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (2):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Lebanon, New Hampshire
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Utrecht
- GSK Investigational Site, Seoul, South Korea

REFERENCES:
- See also: Results for study SKF104864/722 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/SKF104864/722?search=study&study_ids=SKF104864%2F722#rs